CLINICAL TRIAL: NCT05253703
Title: Enhancing Exercise Intensity, Motivation and Enjoyment for Younger and Older Healthy Adults (VCycle-Competition-HA)
Brief Title: Immersive Virtual Reality Bicycling for Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Judith E Deutsch, PT, PhD, Professor, Department of Rehabilitation & Movement Sciences, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2021002091
Record Dates: First submitted 2022-02-10; First posted 2022-02-24 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: competition; exercise; bicycling; aging; virtual reality
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Bicycling (Other): This is a single arm study in which all participants will execute the same three bicycling tasks over one session. Exercise intensity and enjoyment are measured while participants bicycle in a virtual reality environment (wearing virtual reality goggles) in three different conditions lasting approximately 5 minutes each.
  Interventions: Other: Virtual reality bicycling

INTERVENTIONS:
Other: Virtual reality bicycling — This is a single arm study in which all participants will execute the same three bicycling tasks over one session (see arm/group description).

SUMMARY:
This study has four objectives about healthy younger and older adults during immersive virtual reality bicycling:

Determine the effect of visual feedback and competition for younger healthy adults during virtual bicycling on user experience, motivation, enjoyment, perception of effort, and neuromuscular and cardiovascular intensity

Determine the effect of visual feedback and competition for older healthy adults during virtual bicycling on user experience, motivation, enjoyment, perception of effort, and neuromuscular and cardiovascular intensity

Compare younger and older during visual feedback and competition bicycling in terms of: user experience, motivation, enjoyment, perception of effort, neuromuscular and cardiovascular intensity

Determine if attention differs in visual feedback bicycling compared to competition bicycling for younger and older healthy adults

DETAILED DESCRIPTION:
Participants will attend one session lasting about 1.5 hours. They will complete a competitiveness assessment and a questionnaire about physical activity. They will then exercise in three different virtual reality augmented bicycling conditions while wearing a head mounted display (goggles). Each of the three conditions will last approximately 5 minutes and will be followed by questionnaires about the participant's experience.

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years old,
* Able to ride a stationary upright bicycle,
* Able to sign informed consent.

Exclusion Criteria:

* Have a recent history of severe heart disease, severe lung disease, uncontrolled diabetes, traumatic brain injury or any other neurological disorder
* Are unable to follow directions or sign a consent form,
* Do not have adequate vision or hearing ability to see or hear a television,
* Have unstable medical condition or musculoskeletal disorder such as severe arthritis, recent knee surgery, hip surgery, or any other condition that the investigators determine would impair the ability to ride the bicycle,
* Have any other medical condition that prevents bicycling,
* Have moderate depression (score of 10 or more on PHQ-9 screening tool)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Neuromuscular Intensity (Bicycling cadence, revolutions per minute) - Feedback | Session 1 - During the 5-minute feedback bout
  Bicycling cadence collected continuously (1 value per second, 1 Hz)
Neuromuscular Intensity (Bicycling cadence, revolutions per minute) - Self-Competition | Session 1 - During the 5-minute self-competition bout
  Bicycling cadence collected continuously (1 value per second, 1 Hz)
Neuromuscular Intensity (Bicycling cadence, revolutions per minute) - Other-Competition | Session 1 - During the 5-minute other-competition bout
  Bicycling cadence collected continuously (1 value per second, 1 Hz)
Motivation (Intrinsic Motivation Inventory) - Feedback | Session 1 - Immediately after completing the 5-minute feedback bout
  Intrinsic Motivation Inventory - enjoyment, competence, effort, and value subscales (16 questions total). Scores in each subscale are averaged, with a minimum score of 1 and a maximum score of 7. Higher scores indicate higher motivation.
Motivation (Intrinsic Motivation Inventory) - Self-Competition | Session 1 - Immediately after completing the 5-minute self-competition bout
  Intrinsic Motivation Inventory - enjoyment, competence, effort, and value subscales (16 questions total). Scores in each subscale are averaged, with a minimum score of 1 and a maximum score of 7. Higher scores indicate higher motivation.
Motivation (Intrinsic Motivation Inventory) - Other-Competition | Session 1 - Immediately after completing the 5-minute other-competition bout
  Intrinsic Motivation Inventory - enjoyment, competence, effort, and value subscales (16 questions total). Scores in each subscale are averaged, with a minimum score of 1 and a maximum score of 7. Higher scores indicate higher motivation.
Cardiovascular Intensity (Heart rate, beats per minute) - Feedback | Session 1 - During the 5-minute feedback bout
  Heart rate collected continuously (1 value per second, 1 Hz)
Cardiovascular Intensity (Heart rate, beats per minute) - Self-Competition | Session 1 - During the 5-minute self-competition bout
  Heart rate collected continuously (1 value per second, 1 Hz)
Cardiovascular Intensity (Heart rate, beats per minute) - Other-Competition | Session 1 - During the 5-minute other-competition bout
  Heart rate collected continuously (1 value per second, 1 Hz)
Visual Attention (infrared eye-tracking data representing gaze positions in a 3D coordinate plane to be used in calculating dwell time in regions of interest in the virtual simulation) - Feedback | Session 1 - During the 5-minute feedback bout
  3D gaze positions measured continuously (50 values per second, 50 Hz)
Visual Attention (infrared eye-tracking data representing gaze positions in a 3D coordinate plane to be used in calculating dwell time in regions of interest in the virtual simulation) - Self-Competition | Session 1 - During the 5-minute self-competition bout
  3D gaze positions measured continuously (50 values per second, 50 Hz)
Visual Attention (infrared eye-tracking data representing gaze positions in a 3D coordinate plane to be used in calculating dwell time in regions of interest in the virtual simulation) - Other-Competition | Session 1 - During the 5-minute other-competition bout
  3D gaze positions measured continuously (50 values per second, 50 Hz)

SECONDARY OUTCOMES:
Rating of Perceived Exertion - Feedback (start) | Session 1 - Immediately at the start (0-minute mark) of the 5-minute feedback bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Feedback (middle) | Session 1 - At the midpoint (2.5-minute mark) of the 5-minute feedback bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Feedback (end) | Session 1 - At the endpoint (5-minute mark) of the 5-minute feedback bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Self-Competition (start) | Session 1 - Immediately at the start (0-minute mark) of the 5-minute self-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Self-Competition (middle) | Session 1 -At the midpoint (2.5-minute mark) of the 5-minute self-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Self-Competition (end) | Session 1 -At the end (5-minute mark) of the 5-minute self-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Other-Competition (start) | Session 1 -Immediately at the start (0-minute mark) of the 5-minute other-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Other-Competition (middle) | Session 1 -At the midpoint (2.5-minute mark) of the 5-minute other-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Rating of Perceived Exertion - Other-Competition (end) | Session 1 -At the end (5-minute mark) of the 5-minute other-competition bout
  Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Competitiveness (Multidimensional Competitive Orientation Inventory) | Session 1 - Collected once at start of session
  Measured once using the Multidimensional Competitive Orientation Inventory consisting of 12 items from 4 subscales (hyper competitive, self-developmental, anxious, lack of interest) For each subscale, mean scores range from 1-6 with higher scores representing higher levels of that subscale metric.
Ranking of Perceived Effort | Session 1 - once at the end of the session. Collected upon study completion, immediately after finishing the final bicycling condition
  Once, after completing all 3 bicycling conditions, participants will be asked in which of the 3 bicycling conditions they felt they worked the hardest. They will rank the 3 conditions with a score from 1-3, with a 1 indicating the condition in which they felt they worked the hardest and a 3 indicating the condition in which they felt they worked the least hard.
Ranking of Enjoyment | Session 1 - once at the end of the session. Collected upon study completion, immediately after finishing the final bicycling condition
  Once, after completing all 3 bicycling conditions, participants will be asked which of the 3 bicycling conditions they liked the best. They will rank the 3 conditions with a score from 1-3, with a 1 indicating the condition they liked the best and a 3 indicating the condition they liked the least.
Audio recordings of exercise experience | Session 1 - once at the end of the session. Collected upon study completion, immediately after finishing the final bicycling condition
  Once, after completing all 3 bicycling conditions, participants will be asked about their exercise experience. Their responses will be audio recorded to be coded and analyzed qualitatively for themes.

OTHER OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Collected once at start of the session
  The IPAQ is a 27-item questionnaire to measure levels of physical activity. There are 4 main domains of physical activity related to: occupation, transportation, housework, leisure activity. Scores range from 0-19,278 with higher scores representing higher levels of physical activity over the past 7 days.
Patient Health Questionnaire (PHQ-9) | Collected once during screening
  The PHQ-9 is a 9-item questionnaire to rate depression (scored from 0-27 with a lower score indicating lower levels of depression).

CONTACTS AND LOCATIONS:
Overall Officials: Judith E Deutsch, Principal Investigator — Rutgers School of Health Professions
Locations (1):
- Rutgers School of Health Professions, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Immediately following completion of the proposed study, the investigators will submit a de-identified data set of the protocol and links to published papers.
Supporting Information: Study Protocol
Time Frame: The investigators will make study data available immediately following completion.
Access Criteria: Open Access

REFERENCES:
- [Derived] Palmieri JL, Deutsch JE. The effects of competition on exercise intensity and the user experience of exercise, during virtual reality bicycling for healthy adults across the lifespan. BMC Sports Sci Med Rehabil. 2025 Aug 8;17(1):228. doi: 10.1186/s13102-025-01253-9. PMID 40781343

DOCUMENTS (1):
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05253703/ICF_000.pdf